CLINICAL TRIAL: NCT02064907
Title: A Phase 1, Randomized, Open-Label, Single Center, Multiple-Dose, Two-Period, Crossover Study to Assess the Bioavailability, Safety, and Pharmacodynamics of Two 30 mg Dexlansoprazole Delayed-Release Orally Disintegrating Tablets Administered on the Tongue Relative to Oral Administration of One 60 mg Dexlansoprazole Delayed-Release Capsule in Healthy Subjects
Brief Title: Bioavailability, Safety, and Pharmacodynamics of Dexlansoprazole Delayed-Release Orally Disintegrating Tablets in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-390MR(OD)_104; U1111-1151-7112 (Other: World Health Organization)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Bioavailability
Keywords: Drug therapy
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexlansoprazole OD Tablets + Dexlansoprazole Capsules (Experimental): Two Dexlansoprazole 30 mg, delayed-release orally disintegrating tablets, orally, once daily for 5 days in Period 1, followed by a 7 day washout period, followed by one dexlansoprazole 60 mg, capsule, orally, once daily for 5 days in Period 2.
  Interventions: Drug: Dexlansoprazole Delayed Release Orally Disintegrating Tablets; Drug: Dexlansoprazole Delayed Release Capsules
- Dexlansoprazole Capsules + Dexlansoprazole OD (Experimental): Dexlansoprazole 60 mg, capsules, orally, once daily for 5 days in Period 1, followed by a 7 day washout period, followed by two dexlansoprazole 30 mg, delayed-release orally disintegrating tablets, orally, once daily for 5 days in Period 2.
  Interventions: Drug: Dexlansoprazole Delayed Release Orally Disintegrating Tablets; Drug: Dexlansoprazole Delayed Release Capsules

INTERVENTIONS:
Drug: Dexlansoprazole Delayed Release Orally Disintegrating Tablets — Dexlansoprazole delayed-release, orally disintegrating (OD) tablets
Drug: Dexlansoprazole Delayed Release Capsules — Dexlansoprazole delayed-release capsules
  Other Names: Dexilant

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) and Pharmacodynamics (PD) of dexlansoprazole delayed-release orally disintegrating (OD) tablets administered on the tongue and swallowed without water.

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. Dexlansoprazole is being tested to see if two different forms of the medication react the same way in the human body. This study will look at biological samples from people who take an orally disintegrating tablet of dexlansoprazole compared to a swallowed capsule of dexlansoprazole.

The study will enroll approximately 52 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups. Both treatment groups will receive both forms of dexlansoprazole at different time periods:

* Two dexlansoprazole 30 mg orally disintegrating tablets for 5 days
* One dexlansoprazole 60 mg capsule for 5 days.

All participants will be asked to take two tablets or one capsule at the same time each day throughout each treatment period of the study.

This single-centre trial will be conducted in the United States. Participants will make 3 visits to the clinic including two 6-day periods of confinement to the clinic, and will be contacted by telephone 5 to 10 days after last dose of study drug for a follow-up assessment.

The overall time to participate in this study is up to 57 days.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a healthy adult male or female participant by Check-in (Day -1 of Period 1).
4. Is aged 18 to 55 years inclusive, by Screening and the first dosing day (Day 1 of Period 1).
5. Weighs at least 50 kg and has a body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive at Screening.
6. If a male participant is nonsterilized and sexually active with a female partner of childbearing potential, he agrees to use adequate contraception from signing of informed consent form throughout the duration of the study and for 30 days after the last dose of study drug.
7. If a female participant of childbearing potential is sexually active with a nonsterilized male partner, she agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days following the last dose of study drug. Female participants of childbearing potential must have a negative serum pregnancy test at Screening and Check-in (Day -1 of Period 1) and they must not be nursing.
8. Is in good health as determined by a physician based on medical history, vital signs, electrocardiogram (ECG) and physical examination findings at Screening and Check-in (Day -1 of Period 1), as applicable.
9. Has clinical chemistry, hematology, and complete urinalysis (fasted for at least 10 hours) at Screening and Check-in (Day -1 of Period 1) results within the reference range for the testing laboratory unless the out of range results are deemed not clinically significant by the investigator.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Check-in (Day -1 of Period 1).
2. Has ever received dexlansoprazole in a previous clinical study or has received dexlansoprazole or lansoprazole as a therapeutic agent within 28 days prior to Check-in (Day -1 of Period 1).
3. Is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant hematologic, neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine, psychiatric disorder or other abnormality (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of dexlansoprazole delayed-release orally disintegrating (OD) tablets or participant has a known hypersensitivity to any component of the formulation of dexlansoprazole delayed-release capsules or other drug with the same mechanism of action (including esomeprazole, lansoprazole, omeprazole, pantoprazole, or rabeprazole).
6. Consumed alcohol or drugs of abuse within 7 days prior to check-in (Day -1 of Period 1), has a positive test result for alcohol or drugs of abuse at Screening or Check-in (Day -1 of Period 1), or is unwilling to abstain from alcohol and drugs of abuse throughout the study.
7. Has received any known hepatic or renal clearance altering agents (eg, erythromycin, cimetidine, barbiturates, phenothiazines, fluvoxamine, etc.) within 28 days prior to Day -1 of Period 1.
8. Has had an acute, clinically significant illness within 30 days prior to Day 1 of Period 1.
9. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as alcohol consumption exceeding 14 units per week) within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
10. With the exception of acetaminophen, the participant has taken any excluded medication, supplements or food products.
11. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
12. If male, the participant intends to impregnate others or donate sperm during the course of this study or for 30 days thereafter.
13. Has consumed any products containing caffeine and/or xanthine within 72 hours prior to Check-in (Day -1 of Period 1) or is unwilling to abstain from these products for the duration of the study.
14. Has current or recent (within 6 months of screening) gastrointestinal disease including esophageal reflux, frequent (more than once per week) occurrence of heartburn, history of malabsorption (ie, celiac disease, biliary atresia, cholestasis), peptic ulcer disease, or any surgical intervention [eg, cholecystectomy, gastric bypass), which would be expected to influence the absorption of drugs.
15. Has a history of cancer, except basal cell carcinoma of the skin that has not been in remission for at least 5 years prior to Day 1 of Period 1.
16. Has a positive test result for hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV), at Screening or a known history of human immunodeficiency virus infection.
17. Used any nicotine-containing products (including but not limited to cigarettes, pipe, cigar, chewing tobacco, nicotine patch, or nicotine gum) within 28 days prior to Check-in (Day -1 of Period 1), or has a positive cotinine test at Screening or Check-in (Day -1 of Period 1) or is unwilling to abstain from these products for the duration of the study.
18. Has poor peripheral venous access.
19. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 56 days prior to Day 1 of Period 1.
20. Has a Screening or Check-in (Day -1 of Period 1) abnormal (clinically significant) ECG. Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator or medically qualified sub-investigator.
21. Has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: creatinine >1.5 mg/dL, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2.5× the upper limit of normal (ULN), or total bilirubin >2.0 mg/dL.
22. Has a positive breath test result for H pylori at Screening.
23. Has a history of a disorder in metabolizing phenylalanine (phenylketonuria).
24. Cannot tolerate placement of the pH probe.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study from 31 January 2014 (Date first informed consent signed) to 24 April 2014.
Pre-assignment Details: A total of 52 healthy adult participants took part in this study at a single site in the US.
Groups:
- Dexlansoprazole Capsules + Dexlansoprazole OD Tablets: Dexlansoprazole 60 mg, capsules, orally, once daily for 5 days in Period 1, followed by a 7 day washout period, followed by two dexlansoprazole 30 mg, delayed-release orally disintegrating tablets, orally, once daily for 5 days in Period 2.
Period: Period 1
Arm/Group | Dexlansoprazole OD Tablets + Dexlansoprazole Capsules | Dexlansoprazole Capsules + Dexlansoprazole OD Tablets
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Dexlansoprazole OD Tablets + Dexlansoprazole Capsules | Dexlansoprazole Capsules + Dexlansoprazole OD Tablets
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population consisted of all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole OD Tablets + Dexlansoprazole Capsules | Dexlansoprazole Capsules + Dexlansoprazole OD Tablets | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (10.11) | 39.1 (10.70) | 37.6 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 19 | 13 | 32
  Non-Hispanic or Latino | 7 | 13 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 24 | 49
  Black/African American | 1 | 2 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.92 (2.540) | 26.44 (2.274) | 26.18 (2.401)
Smoking classification [Number; unit: participants]
  Never smoked | 25 | 17 | 42
  Current smoker | 0 | 0 | 0
  Ex-smoker | 1 | 9 | 10
Alcohol classification [Number; unit: participants]
  Has never drunk | 18 | 16 | 34
  Current drinker | 6 | 6 | 12
  Ex-drinker | 2 | 4 | 6
Caffeine consumption [Number; unit: participants]
  Yes | 6 | 9 | 15
  No | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Dexlansoprazole on Day 1.
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 predose and up to 24 hours post-dose
Population: Participants from the PK population - all participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration-with data available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dexlansoprazole OD Tablets: Two dexlansoprazole 30 mg, delayed-release orally disintegrating tablets, orally, once daily for 5 days.
- Dexlansoprazole Capsules: Dexlansoprazole 60 mg, capsules, orally, once daily for 5 days.
Arm/Group | Dexlansoprazole OD Tablets | Dexlansoprazole Capsules
Number analyzed (Participants) | 52 | 52
ng/mL | 1046.8846 (496.79560) | 1164.3654 (667.01483)

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Dexlansoprazole on Day 5
Description: as for outcome 1
Time Frame: Day 5 predose and up to 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dexlansoprazole OD Tablets | Dexlansoprazole Capsules
Number analyzed (Participants) | 52 | 52
ng/mL | 1150.8462 (668.54581) | 1178.1346 (570.01221)

3. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration on Day 1
Description: AUC(0-tlqc) is a measure of total plasma exposure to a drug from time 0 to time of the last quantifiable concentration.
Time Frame: Day 1 predose and up to 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dexlansoprazole OD Tablets | Dexlansoprazole Capsules
Number analyzed (Participants) | 52 | 52
ng*hr/mL | 5059.5689 (3689.92045) | 6746.6075 (5489.74215)

4. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration on Day 5
Description: AUC(0-tlqc) is a measure of total plasma exposure to a drug from time 0 to time of the last quantifiable concentration.
Time Frame: Day 5 predose and up to 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dexlansoprazole OD Tablets | Dexlansoprazole Capsules
Number analyzed (Participants) | 52 | 52
ng*hr/mL | 5818.8236 (5105.56325) | 7184.1729 (6313.98668)

5. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity on Day 1
Description: AUC(0-inf) is a measure of the area under the plasma concentration-time curve from time 0 extrapolated to infinity.
Time Frame: Day 1 predose and up to 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dexlansoprazole OD Tablets | Dexlansoprazole Capsules
Number analyzed (Participants) | 52 | 50
ng*hr/mL | 5364.0217 (4218.37276) | 7155.4994 (6461.07333)

6. Primary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval on Day 5
Description: AUC(0-tau) is a measure of the area under the plasma concentration-time curve from time 0 to time tau over a dosing interval, where tau is the length of the dosing interval (24 hours).
Time Frame: Day 5 predose and up to 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dexlansoprazole OD Tablets | Dexlansoprazole Capsules
Number analyzed (Participants) | 52 | 52
ng*hr/mL | 5824.7108 (5105.49002) | 7196.1922 (6306.70574)

ADVERSE EVENTS:
Time Frame: From first dose date up to 30 days from the last dose date
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dexlansoprazole OD Tablets | Dexlansoprazole Capsules
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 10/52 | 12/52
OTHER ADVERSE EVENTS (reported when occurring in more than 3.8% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole OD Tablets (N=52) | Dexlansoprazole Capsules (N=52)
Nausea (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2
Headache (Nervous system disorders) | 5 | 6
Dizziness (Nervous system disorders) | 2 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property